CLINICAL TRIAL: NCT02377882
Title: The Optimal Dosage of Neuromuscular Blocking Agent for Intraoperative Neuromonitoring During Thyroid Surgery
Brief Title: The Optimal Dosage of Rocuronium for Intraoperative Neuromonitoring During Thyroid Surgery
Acronym: IONM
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Koung-Shin Chu, visiting staff, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-980170
Record Dates: First submitted 2010-07-08; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: THYROIDECTOMY
Keywords: Intra-operative neuromonitoring; Neuromuscular blocking agent; Rocuronium; Thyroid surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators tried to explore an alternative non-depolarizing muscle relaxant (rocuronium) and its optimal dosage to replace succinylcholine for IONM during thyroid surgery.Time frame of outcome measure was during 30 to 70min after rocuronium injection. Specific time points at which the will be assessed and for EMG signals will be presented.

DETAILED DESCRIPTION:
Recurrent laryngeal nerve (RLN) palsy is the most common and serious complication after thyroid surgery, and ranks among the leading reasons for medicolegal litigation of surgeons. Intraoperative neuromonitoring (IONM) are being applied to prevent RLN injury during thyroid surgery. IONM has been used as a means not only to localize and identify the RLN, but also to predict cord function and elucidate the surgical pitfalls during preparation of RLN.

Muscle relaxant is necessary for general anesthesia; it can facilitate tracheal intubation and stable conditions for surgery. However, the use of muscle relaxant might diminish the EMG response during IONM and interfere with the interpretation of IONM results. Eighty patients were randomized to receive one (group 1, n=40) or two (group 2, n=40) effective dose (ED95) of rocuronium to facilitate EMG endotracheal tube insertion. Evoked potentials were obtained per 5 minutes by stimulating vagus nerve from the time point of 30 to 70 minutes after administration of rocuronium. The magnitude of evoked potential at each time point and tracheal intubating condition were compared between groups. Accelerometry [twitch (% TW)] was used to monitor the quantitative degree of neuromuscular transmission. The aim of this study was to explore an alternative non-depolarizing muscle relaxant (Rocuronium) and its optimal dosage to replace succinylcholine for IONM. The ED95 of rocuronium is 0.3mg/kg and 2×ED95 is generally recommended as a standard intubation dosage.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of thyroid tumor

Exclusion Criteria:

* neuromuscular disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were planned to receive thyroidectomy
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The time to detect V1 and V2 signals | WITHIN 2 DAYS, follow up to 6 months
  V1 signal means an EMG signals obtained from the vagus nerve before identification of RLN.
  V2 signal-The final testing of the vagus nerve EMG signals was performed after complete hemostasis of the operative field.
  The amplitude (μV) of V1 and V2 signals and the correlated degree of neuromuscular transmission (% TW) were recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: I-Chen Lu, M.D., Study Chair — Department of Anesthesiology, Kaohsiung Medical University Hospital, Kaohsiung Medical University, Kaohsiung, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Dralle H, Sekulla C, Lorenz K, Brauckhoff M, Machens A; German IONM Study Group. Intraoperative monitoring of the recurrent laryngeal nerve in thyroid surgery. World J Surg. 2008 Jul;32(7):1358-66. doi: 10.1007/s00268-008-9483-2. PMID 18305996
- [Background] Chan WF, Lo CY. Pitfalls of intraoperative neuromonitoring for predicting postoperative recurrent laryngeal nerve function during thyroidectomy. World J Surg. 2006 May;30(5):806-12. doi: 10.1007/s00268-005-0355-8. PMID 16680596
- [Background] Chan WF, Lang BH, Lo CY. The role of intraoperative neuromonitoring of recurrent laryngeal nerve during thyroidectomy: a comparative study on 1000 nerves at risk. Surgery. 2006 Dec;140(6):866-72; discussion 872-3. doi: 10.1016/j.surg.2006.07.017. Epub 2006 Sep 18. PMID 17188132